CLINICAL TRIAL: NCT03206762
Title: JETStream AtheRectomy With Adjunctive Paclitaxel-Coated BallooN Angioplasty vs Balloon AnGioplasty Followed by Paclitaxel-Coated Balloon in Treating ComplEx Denovo FemoRopopliteal Arterial Disease (JET-RANGER)
Brief Title: JET-RANGER Trial - JETStream Atherectomy With Adjunctive Paclitaxel-Coated Balloon Angioplasty vs Plain Old Balloon Angioplasty Followed by Paclitaxel-Coated Balloon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Cardiovascular Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCRF-S-001-2015
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: 255 subjects are planned for enrollment (with a block 2:1 randomization)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Jetstream Atherectomy+Ranger DCB or Medtronic IN.PACT DCB (Experimental): Jetstream Atherectomy used in conjunction with the Ranger DCB or Medtronic IN.PACT DCB
  Interventions: Device: Jetstream Atherectomy with randomization to the Ranger or IN.PACT DCB Arm or the POBA+DCB (Ranger or IN.PACT) Arm
- POBA+DCB (Ranger or IN.PACT) (Active Comparator): POBA and then DCB treatment (Ranger or IN.PACT)
  Interventions: Device: Jetstream Atherectomy with randomization to the Ranger or IN.PACT DCB Arm or the POBA+DCB (Ranger or IN.PACT) Arm

INTERVENTIONS:
Device: Jetstream Atherectomy with randomization to the Ranger or IN.PACT DCB Arm or the POBA+DCB (Ranger or IN.PACT) Arm — Jetstream Atherectomy with randomization to the Ranger or IN.PACT DCB Arm or the POBA+DCB (Ranger or IN.PACT) Arm

SUMMARY:
A prospective, multicenter, randomized study evaluating the use of Jetstream Atherectomy (JS) followed by DCB in comparison to the use of plain old balloon angioplasty (POBA) followed by DCB alone in the treatment of complex lesions in femoropopliteal arteries in subjects with claudication (Rutherford Clinical Category (RCC) of 2-4) (complex lesions are defined as long (≥ 10 cm) lesions, or moderately or highly calcified lesions, or chronic total occlusions irrespective of length).

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following general inclusion criteria.

1. Has a Rutherford Clinical Category of 2 - 4.
2. Is willing and capable of complying with all follow-up evaluations at the specified times (including an angiogram at the 1-year follow-up visit).
3. Is ≥ 18 years old.
4. Is able and willing to provide written informed consent prior to study specific procedures.

Angiographic Inclusion Criteria:

Subject must meet all of the following angiographic inclusion criteria. Unless otherwise specified, the Investigator performing the procedure bases all angiographic inclusion criteria on visual determination at the time of the procedure.

1. Has evidence at the target lesion of ≥ 70% de novo stenosis of a. ≥ 10 cm length, or b. any chronic total occlusion (> 1 month by history or known by conventional or CT angiography or arterial duplex ultrasound) in the SFA (at least 1 cm from the bifurcation of the profunda) and/or popliteal artery, or 3. at least grade 2 or higher calcification as defined by the peripheral arterial calcium scoring system (PACCS)26
2. Has evidence of at least one runoff vessel to the ankle/foot of the limb to be treated that does not have significant (< 70%) stenosis during the index procedure.
3. Has a reference vessel diameter of 4 - 7 mm.
4. Has a target lesion an exchangeable guidewire can cross via the true lumen (without using a re-entry device or a subintimal approach).

General Exclusion Criteria:

The subject must not meet any of the following general exclusion criteria.

1. Has one or more of the contraindications listed in the JetStream or Ranger IFUs.
2. Has a contraindication or known untreated allergy to antiplatelet therapy, anticoagulants, thrombolytic drugs or any other drug anticipated to be used (that cannot be reasonably substituted).
3. Is expected to require cilostazol (Pletal) during the one-year follow-up period.
4. Has a hypersensitivity to contrast material that cannot be adequately pretreated.
5. Has known hypersensitivity to treatment device materials including paclitaxel or nitinol.
6. Has known uncontrollable hypercoagulable condition, or refuses blood transfusion.
7. Has life expectancy of less than 24 months.
8. Is pregnant, of childbearing potential not taking adequate contraceptive measures, or nursing.
9. Has surgical or endovascular procedure of the target vessel within 30 days prior to the index procedure.
10. Has any planned surgical intervention (requiring hospitalization) or endovascular procedure within 30 days after the index procedure.
11. Is currently participating in an investigational drug or another device study that may clinically interfere with the study outcomes.
12. Has any co-morbid condition that in the judgment of the physician precludes safe percutaneous intervention.
13. Has had a previous peripheral bypass affecting the target vessel (allowable for physician to pass through bypass graft in aorta-iliac region to get to the target lesion).
14. Has chronic renal insufficiency (eGFR < 30 ml/min or creatinine ≥ 2.5 including dialysis patients).
15. Has planned laser, cryo, TurboHawk or any other treatment except study treatment within 30 days after the index procedure.
16. Has had superficial thrombophlebitis or deep venous thrombus within 30 days prior to index procedure.
17. Has had a stroke within 3 months prior to index procedure.
18. Has had a myocardial infarction within 1 month prior to index hospitalization
19. Has history of significant gastrointestinal bleeding in the past 2 months prior to index procedure, or any history of hemorrhagic diathesis.
20. Has a known or suspected systemic infection at the time of the index procedure.
21. Patients with ipsilateral Iliac and CFA disease are allowed in the study but these lesions have to be treated successfully first (<30% residual) before patient can be enrolled. Treatment as per investigator's preference.
22. Aneurysm located in the target vessel or aneurysmal vessel

Angiographic Exclusion Criteria:

The subject must not meet any of the following angiographic exclusion criteria. The Investigator performing the procedure bases all angiographic exclusion criteria on visual determination at the time of the procedure.

1. Has < 70% stenosis prior to treatment of the target lesion.
2. Has in-stent restenosis of the target lesion.
3. Has an acute intraluminal thrombus within the target lesion.
4. Has an aneurysmal target vessel
5. Patient has already been enrolled in the study or any other study that by the investigator judgment may interfere with the outcome of this trial
6. Has two or more lesions that require treatment in the target vessel. Lesions have to be separated by > 5 cm in order to be considered different lesions. Only one lesion per target vessel can be enrolled during the index procedure
7. Has disease that precludes safe advancement of the JS device to the target lesion.
8. P3 segments of the popliteal vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Target Lesion Revascularization | 1 year
  Effectiveness: Target Lesion Revascularization at 1 Year: TLR is defined as retreatment of the index lesion (extended 1 cm proximal and distal to the lesion) at 1 year. For the primary endpoint, intra-procedural bail out stenting of the index lesion is considered meeting a TLR endpoint. (ITT analysis)
Major Adverse Events | 30 Days
  Safety: Major Adverse Events (MAE) at 30 days: unplanned amputation, total mortality or TLR at 30 days (TLR includes bail out stenting)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Shammas, MD, Research Director, Study Director — MCRF
Locations (1):
- Midwest Cardiovascular Research Foundation, Davenport, Iowa, United States